CLINICAL TRIAL: NCT01845155
Title: Neuro-Music-Therapy for Patients With Chronic Tinnitus - a Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Center for Music Therapy Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMTR-TC-02
Record Dates: First submitted 2013-04-24; First posted 2013-05-03 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Tinnitus
Keywords: Tinnitus; music therapy; directive counselling; acoustic stimulation; group comparison; subjective evaluation; pitch
MeSH Terms: conditions — Tinnitus | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Music Therapy (Experimental): Neuro-Music-Therapy according to the Heidelberg Model
  Interventions: Behavioral: Neuro-Music-Therapy according to the Heidelberg Model
- Counselling (Active Comparator): Counselling
  Interventions: Behavioral: Counselling

INTERVENTIONS:
Behavioral: Neuro-Music-Therapy according to the Heidelberg Model — The neuro-music therapy according to the Heidelberg Model for tinnitus is a manualized short term music therapeutic treatment lasting for nine consecutive 50-minutes sessions of individualized therapy. Therapy takes place on five consecutive days (from Monday to Friday) with two therapy sessions per day. It comprises both active and receptive forms of music therapy. The interventions are structured into the following modules Directive Counseling, Resonance Training, Neuroauditive Cortex Training, Tinnitus Reconditioning.
  For more details on the music therapy see Argstatter et al. 2012
  Arms: Music Therapy
Behavioral: Counselling — Duration: single session of 50 min Tinnitus specific procedures: The counseling group receives the identical counselling procedure as the music therapy group.
  Arms: Counselling

SUMMARY:
BACKGROUND: Tinnitus is a nonspecific symptom of hearing disorder characterized by the sensation of buzzing, ringing, clicking, pulsations, and other noises in the ear. Despite a variety of treatments, many patients with chronic tinnitus ask for more active ways in coping with their tinnitus. Gold standard treatment in chronic tinnitus is a comprehensive directive counseling explaining the underlying mechanisms leading to the tinnitus percept. Therefore a neuro-music therapeutic treatment based on a bio-psycho-social framework was developed and compared to a counselling-only control group.

INTERVENTION: two standardized protocols for tinnitus therapy were defined ("neuro-music therapy" vs. "counselling")

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic tinnitus persisting for a minimum of 6 month
* Adults, aged 18 or over
* Patients are able to understand, read and speak German fluently
* Patients are able to give written informed consent
* tinnitus with determinable centre frequency

Exclusion Criteria:

* Tinnitus related to anatomic lesions of the ear, to retrocochlear lesions or to cochlear implantation
* Tinnitus is concomitant symptom of a known systemic disease (such as Menière's Disease, vestibular schwannoma, endolymphatic hydrops)
* Status following craniocerebral trauma, cervicogenic or stomatognathic tinnitus
* Tinnitus is neither noisiform nor tonal (cricking, clacking, rumbling) or has different sound components or is pulsatile, intermittent or non-persistent
* Severe hearing impairment (greater than 50 decibel hearing loss (dB HL) in the region of the centre tinnitus frequency)
* Severe hyperacusis
* One or two sided deafness
* Clinical diagnosis of severe mental disorder or psychiatric or neurological disease (psychosis, epilepsy, Parkinsons's disease, dementia, alcohol or drug abuse)
* History of severe ischemic disorder (previous stoke, previous heart attack, peripheral arterial occlusion disease)
* Inability to discontinue drugs known to be associated with tinnitus (high-dose aspirin, quinidine, aminoglycosides) or psychotropic medication prior to entry into the study
* Patients are not able to understand, read and speak German fluently
* Patients are not able to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-03; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heike Argstatter, Dr, Principal Investigator — German Center for Music Therapy Research
Locations (1):
- German Center for Music Therapy Research, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Argstatter H, Grapp M, Hutter E, Plinkert P, Bolay HV. Long-term effects of the "Heidelberg Model of Music Therapy" in patients with chronic tinnitus. Int J Clin Exp Med. 2012;5(4):273-88. Epub 2012 Aug 22. PMID 22993646
- [Derived] Argstatter H, Grapp M, Hutter E, Plinkert PK, Bolay HV. The effectiveness of neuro-music therapy according to the Heidelberg model compared to a single session of educational counseling as treatment for tinnitus: a controlled trial. J Psychosom Res. 2015 Mar;78(3):285-92. doi: 10.1016/j.jpsychores.2014.08.012. Epub 2014 Sep 3. PMID 25224125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was announced by press releases in German leading to self-admittance to the Heidelberg Out-patient Center for Tinnitus. It was offered to patients by ENT-doctors in own practice nationwide and to patients attending the ENT-clinic of the university hospital Heidelberg. Recruitment took place between March 2006 and February 2013.
Pre-assignment Details: complete audiometric and psychological profile (exclusion of 10 patients due to incomplete data)
Groups:
- Music Therapy: Neuro-Music-Therapy according to the Heidelberg Model
  Neuro-Music-Therapy according to the Heidelberg Model : The neuro-music therapy according to the Heidelberg Model for tinnitus is a manualized short term music therapeutic treatment lasting for nine consecutive 50-minutes sessions of individualized therapy. Therapy takes place on five consecutive days (from Monday to Friday) with two therapy sessions per day. It comprises both active and receptive forms of music therapy. The interventions are structured into the following modules Directive Counseling, Resonance Training, Neuroauditive Cortex Training, Tinnitus Reconditioning.
  For more details on the music therapy see Argstatter et al. 2012
- Counselling: Counselling
  Counselling : Duration: single session of 50 min Tinnitus specific procedures: The counseling group receives the identical counselling procedure as the music therapy group.
Period: Overall Study
Arm/Group | Music Therapy | Counselling
Started | 146 | 144
Completed | 145 | 144
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Music Therapy | Counselling | Total
Number analyzed (Participants) | 146 | 144 | 290
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 119 | 244
  >=65 years | 21 | 25 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (11.6) | 53.2 (11.9) | 52.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 96 | 200
  Male | 42 | 48 | 90
Region of Enrollment [Number; unit: participants]
  Germany | 146 | 144 | 290
TQ-score [Mean (Standard Deviation); unit: units on a scale] | 33.0 (14.8) | 32.9 (13.4) | 32.9 (15.0)
Tinnitus Pitch [Mean (Standard Deviation); unit: Hz] | 5805 (2594) | 5851 (2678) | 5834 (2622)

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Questionnaire (TQ, Goebel and Hiller 1998) Total Score Change From Baseline to End of Treatment
Description: Tinnitus severity was assessed by the German version of the tinnitus questionnaire (TQ, Goebel and Hiller 1994). The TQ consists of a total of 52 items. The questionnaire records tinnitus related complaints on a global TQ-score. The range of values is between the minimum score of 0 and the maximum score of 84, whereas high values indicate high tinnitus related distress.
Time Frame: average time period was 3 months
Measure: Mean (Standard Deviation); unit: absolute TF-score change
Arm/Group | Music Therapy | Counselling
Number analyzed (Participants) | 146 | 144
absolute TF-score change | 13.6 (7.4) | 3.7 (6.8)

2. Secondary Outcome: Change in Tinnitus Frequency (Pitch), Obtained at Admission (Pre) and After Therapy Intervention (Post)
Time Frame: the average time period was 3 months
Measure: Median (Standard Deviation); unit: Hz
Arm/Group | Music Therapy | Counselling
Number analyzed (Participants) | 146 | 144
Hz | 2342 (3768) | 530 (2036)

ADVERSE EVENTS:
Arm/Group | Music Therapy | Counselling
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes